CLINICAL TRIAL: NCT07244497
Title: Evaluation of a Dementia Communication Training Program Using a Real-time Interactive Virtual Trainer Among Novice Home Care Workers
Brief Title: Dementia Communication Training Program for Novice Home Care Workers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tzu Chi University (Other)
Responsible Party: Principal Investigator, Huei-Chuan Sung, Associate professor, Tzu Chi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: YLH-IRB-11326
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Dementia
Keywords: virtual technology; dementia; communication skill; novice home care worker
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Masking Description: Data assessors will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual trainer-based dementia communication training (Experimental): 8-week dementia communication training program using a real-time interactive virtual trainer
  Interventions: Other: virtual trainer-based dementia communication training
- scenario-based discussions dementia communication training (Active Comparator): 8-week dementia communication training program using scenario-based discussions
  Interventions: Other: scenario-based discussions dementia communication training

INTERVENTIONS:
Other: virtual trainer-based dementia communication training — 8-week dementia communication training program using a real-time interactive virtual trainer
  Arms: virtual trainer-based dementia communication training
Other: scenario-based discussions dementia communication training — 8-week dementia communication training program using scenario-based discussions
  Arms: scenario-based discussions dementia communication training

SUMMARY:
This study aims to evaluate the effects of a dementia communication training program using a real-time interactive virtual trainer among novice home care workers.

DETAILED DESCRIPTION:
This randomised controlled trial aims to evaluate the effects of a dementia communication training program using a real-time interactive virtual trainer on dementia knowledge, communication skills, empathy, and competence of managing behavioral and psychological symptoms of dementia (BPSD) among novice home care workers.

The virtual trainer (VT) group will receive the 8-week virtual trainer-based dementia communication training.

The control group will receive the 8-week scenario-based discussions dementia communication training.

Both groups will be assessed for their dementia knowledge, communication skills, empathy, and competence of managing BPSD at baseline, week 4, and week 18, and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Novice home care workers who had been employed in home care agencies for less than one year.
* ages ranging from 20 to 65 years,
* completed care worker training program
* Had not previously received any virtual trainer training.
* Taiwanese nationality
* provided informed consent to participate in the study.

Exclusion Criteria:

* home care workers who do not meet the inclusion criteria

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Dementia Knowledge Assessment Scale | baseline, week 4, week 8, week 12
  Dementia Knowledge, total score ranges from 0 to 50, with higher scores indicating a higher level of knowledge.
Caregiver Communication Competence Scale | baseline, week 4, week 8, week 12
  communication skills, total score ranges from 14 to 56, with higher scores indicating stronger communication skills.

SECONDARY OUTCOMES:
Jefferson Scale of Empathy | baseline, week 4, week 8, week 12
  empathy, total score ranges from 20 to 140, with higher scores indicating a more positive level of empathy.
Competence Scale in Managing Behavioral and Psychological Symptoms of Dementia | baseline, week 4, week 8, week 12
  Competence in Managing Behavioral and Psychological Symptoms of Dementia, the total score ranges from 28 to 140, with higher scores indicating better ability to manage behavioral and psychological symptoms of dementia (BPSD).

CONTACTS AND LOCATIONS:
Overall Officials: HUEICHUAN SUNG, Principal Investigator — Tzu Chi University

IPD SHARING:
Plan to Share IPD: No